CLINICAL TRIAL: NCT05742828
Title: Virtual Seating Coach on Power Wheelchairs of Persons With ALS
Brief Title: Virtual Seating Coach on Power Wheelchairs of Persons With Amyotrophic Lateral Sclerosis (ALS)
Acronym: ALS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Permobil, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00082646
Record Dates: First submitted 2023-02-15; First posted 2023-02-24 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-02

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Power wheelchairs; pressure injuries; pain
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Pressure Ulcer; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Seating Coach (Active Comparator): The Virtual Seating Coach is a context-aware reminding system that when set up by a clinician, directly benefits a user by reminding him or her to change position with the chair's power seating function.. Regular position changes increase independent function, reduce the risk of pressure ulcers, manage pain, and reduce swelling.
  Interventions: Behavioral: Virtual Seating Coach
- Non Virtual Seating Coach (No Intervention): power wheelchairs that tilt, recline, and have leg elevation for maximal pressure management and to encourage repositioning to reduce the risk of skin breakdown/pressure injury as well as decrease pain.

INTERVENTIONS:
Behavioral: Virtual Seating Coach — Power wheelchair intervention
  Arms: Virtual Seating Coach

SUMMARY:
A literature review was completed related to the topic of use of the Virtual Seating Coach (VSC) device with clients with Amyotrophic Lateral Sclerosis (ALS) with no results. The VSC components are FDA approved and Health Insurance Portability and Accountability Act (HIPPA) compliant, which have been used for many years by clinicians to achieve therapy goals of repositioning and best practice of utilizing power wheelchair seat functioning on a frequent basis. The VSC is typically not covered by insurance, but with clinical documentation, it has the potential for reimbursement. There is conflicting and vague information in the literature with regards to the prevalence/types of wounds and prevalence of pain in this population.

DETAILED DESCRIPTION:
According to most literature, clients with ALS in general, get few pressure injuries. At this clinic, however, potentially due to the longer life expectancy of clients who choose tracheostomy with mechanical ventilation and a feeding tube, some clients do get pressure injuries. Also, many clients once they are sitting most of the day, whether in the wheelchair, recliner or bed, complain of discomfort and pain. Most clients will use or require a power wheelchair for mobility and positioning in the course of the disease process, and many will require it full time as symptoms progress. Generally, decreased sensation is not a symptom of ALS, but it is unknown why some people with ALS have pain and pressure injuries despite the intact sensation needed to cue repositioning.

It is best clinical practice to provide clients with ALS power wheelchairs that tilt, recline, and have leg elevation for maximal pressure management and to encourage repositioning to reduce the risk of skin breakdown/pressure injury as well as decrease pain. This study will study the effect of having an alerting/coaching system for training and reminders on performing pressure relief and repositioning for decreasing the number of pressure injuries as well as decreasing pain. The VSC also gives contextual cues to achieve a specific angle set-up by the clinician. Not only does the VSC provide alerts, but the client and clinician can observe and track the amount of time the chair is on and in what position.

ELIGIBILITY:
Inclusion Criteria:

Treatment group:

* Inclusion will be diagnosis of amyotrophic lateral sclerosis (ALS)
* Current clinic client at The Carolinas Neuromuscular ALS/MDA Center's Multidisciplinary ALS clinic
* Currently using a Permobil power wheelchair with power seating with R-Net electronics that accepts the VSC
* Has a Permobil Corpus 3G (6 months old or newer) or who order a new Permobil power wheelchair.
* New Permobil chairs which are not obtained through this clinic will also be able to enter the study, such as chairs from other regions or from the Veteran's Administration.

Comparison group:

* Inclusion will be diagnosis of ALS
* Current clinic client at The Carolinas Neuromuscular ALS/Muscular Dystrophy Association (MDA) Center's multidisciplinary ALS clinic
* Currently using a power wheelchair with power seating.
* New chairs which are not obtained through this clinic will also be able to enter the study, such as chairs from other regions or from the Veteran's Administration.

Exclusion Criteria:

Treatment group:

* Another diagnosis besides ALS
* Does not have a Smart phone or tablet
* Frontotemporal Dementia as noted by MD/SLP/SW (Medical Doctor/Speech Language Pathologist/Social Worker) in medical records
* Inability/unwillingness to control wheelchair power features (client)
* Unwillingness to be monitored by study staff and alerted by VSC over time
* Uses other mobility devices indoors (scooter, basic power wheelchair) more than or in addition to Permobil PWC

Comparison group:

* Another diagnosis besides ALS
* Frontotemporal Dementia as noted by MD/SLP/SW in medical records
* Inability/unwillingness to control wheelchair power features (client)
* Unwillingness to be monitored by study staff
* Uses other mobility devices indoors (scooter, basic power wheelchair) more than or in addition to power wheelchair
* Further exclusions may be added in future protocol versions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Change in seat function utilization with use of the Virtual Seating Coach (VSC) | Year 3
  tracked through the Virtual Seating Coach app and Permobil data collection
Change in number of Complications | Year 3
  Pressure and pain questions measured using a Likert Scale - A type of psychometric response scale in which responders specify their level of agreement to a statement typically in five points: (1) Strongly disagree; (2) Disagree; (3) Neither agree nor disagree; (4) Agree; (5) Strongly agree.

SECONDARY OUTCOMES:
Change in Utilization of VSC | Year 3
  If limitations are addressed (respiratory, cushion, comfort, control) does utilization increase? - evaluated with surveys and phone calls

CONTACTS AND LOCATIONS:
Overall Officials: Amber Ward, MS, OTR/L, Principal Investigator — Carolinas Neuromuscular ALS/MDA Center
Locations (1):
- Atrium Health - Neurosciences Institute, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2017-12-28): https://cdn.clinicaltrials.gov/large-docs/28/NCT05742828/ICF_000.pdf